CLINICAL TRIAL: NCT07396142
Title: Application of BaiXiaoAi Companion AI in the Diagnosis, Treatment, and Follow-up Management of Oncology Patients: A Single-Center, Prospective, Exploratory Study
Brief Title: BaiXiaoAi AI Companion for Cancer Patient Follow-up
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING_LI, Chief, Office of Clinical Trial Center, CancerIHCAMS, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCCH0047
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Symptoms and Signs; Artificial Intelligence; Artificial Intelligence Mobile Application; Needs Assessment
Keywords: WeChat-based AI companion; Tumor patients,; Cancer patients; Patient satisfaction; Symptom management; Emotional support; Clinical needs assessment
MeSH Terms: conditions — Signs and Symptoms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Study Population: This is an observational study with no predefined study groups
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational study. No experimental intervention (including drugs, devices, etc.) will be administered to the participants. The investigators will only collect clinical data and follow-up outcomes of the participants according to the study protocol.

SUMMARY:
This is a prospective, single-center, exploratory study designed to evaluate the accuracy, user engagement, and user experience of the BaiXiaoAi Companion AI. Upon signing the informed consent form and enrollment, a dedicated "Doctor-Nurse-Patient-AI" WeChat group will be established for each participant. Within the group, the BaiXiaoAi AI will provide timely responses based on patient communications and proactively push information regarding disease management and patient education.

DETAILED DESCRIPTION:
This is a prospective, single-center, exploratory clinical study aiming to comprehensively assess the diagnostic accuracy, user engagement efficacy, and subjective user experience of the BaiXiaoAi Companion AI system in the context of clinical patient management.

Following the voluntary signing of the informed consent document and formal enrollment into the study cohort, each participant will be assigned to a dedicated WeChat group adopting a "Doctor-Nurse-Patient-AI" quadruple collaborative model. Within this closed communication platform, the BaiXiaoAi Companion AI is programmed to perform two core functions: first, it delivers real-time, contextually tailored responses to patients' inquiries, symptom descriptions, and daily health-related communications shared within the group; second, it proactively disseminates personalized, evidence-based content covering disease-specific management protocols, medication adherence guidance, lifestyle modification recommendations, and targeted patient education materials. These interventions are designed to facilitate seamless interaction between medical providers and patients while leveraging AI-driven tools to augment the continuity of care outside of traditional clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older;
* Patients with a confirmed diagnosis of malignant neoplasms who are currently undergoing treatment or in follow-up, or their primary caregivers;
* Able to read and communicate in Chinese and independently use WeChat;
* Willing and able to provide informed consent.

Exclusion Criteria:

* Presence of severe psychiatric disorders (e.g., schizophrenia, bipolar disorder) or cognitive impairment (MMSE score < 24);
* Inability to use WeChat or communicate in Chinese;
* Considered by the investigators to be unsuitable for participation due to psychological or physical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with malignant neoplasms who are undergoing cancer treatment or follow-up at a single study center, as well as their primary caregivers. Participants are enrolled after providing informed consent and are followed prospectively for observational data collection related to communication needs and usage patterns during routine care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy and safety of AI-assisted patient communication | Up to 12 months
  The accuracy and safety of the AI-assisted communication tool will be assessed by monitoring the occurrence and severity of AI-related safety events during the study period. Safety events include misinformation, misunderstanding, inappropriate emotional responses, or potential risks related to medical decision-making attributable to the AI tool. Events are classified into four levels (Grade 0-3), where Grade 0 indicates no issue and Grade 3 indicates a serious error with potential medical risk.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences